CLINICAL TRIAL: NCT06334523
Title: Open Randomised Study of Conventional Ventilation Optimised by Dead Space Washout in Extremely Premature Infants
Brief Title: Ventilation of the Extremely Premature Infants Optimized by Dead Space Washout
Acronym: Volem
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Volem
Record Dates: First submitted 2024-03-18; First posted 2024-03-28 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Extremely Low Birthweight Infant; Continuous Tracheal Gas Insufflation; Medical Device; Lung Protection; Ventilator-Induced Lung Injury
Keywords: lung protection; extremely low birthweight infant; Ventilator-Induced Lung Injury; mechanical ventilation
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Continuous Tracheal Gas Insufflation (Experimental): the preterm infant intubated and ventilated with Continuous Tracheal Gas Insufflation
  Interventions: Device: Ventilation with Dead Space Washout via Continuous Tracheal Gas Insufflation (CTGI)
- Standard ventilation without CTGI (No Intervention): In the No Intervention arm, the preterm infants are mechanically ventilated using standard ventilation, without the CTGI-device. There is no dead space washout.

INTERVENTIONS:
Device: Ventilation with Dead Space Washout via Continuous Tracheal Gas Insufflation (CTGI) — The intervention involves adding a device which allows CTGI (the "CTGI-device") to washout the dead space in preterm mechanically ventilated infants. Dead space washout using the CTGI-device is an option added to standard ventilation, to reduce or even cancel anatomical dead space due to respiratory prostheses in intubated preterm infants.
  Other Names: Continuous Tracheal Gas Insufflation; CTGI
  Arms: Continuous Tracheal Gas Insufflation

SUMMARY:
The Continuous Tracheal Gas Insufflation (CTGI) is a ventilation option of conventional mechanical ventilation that is used to reduce or even eliminate the dead space caused by respiratory prostheses. This objective is of particular interest in the smallest preterm infants, where the volume of anatomical dead space due to prostheses is little different from the tidal volume. The principle of this option is to continuously blow an additional flow of 0.2 L/minute at the tip of the endotracheal tube to purge expired CO2 trapped in the prostheses, to have a CO2-free volume of gas available for subsequent insufflation.

The goal of this clinical trial is to learn if Continuous Tracheal Gas Insufflation (CTGI) works to reduce ventilatory dependence in preterm infants after mechanical ventilation. It will also learn about the safety of CTGI. The main questions it aims to answer are:

* Does Continuous Tracheal Gas Insufflation (CTGI) reduce the number of days of non-invasive ventilation in extremely preterm infants who needed mechanical ventilation?
* Does Continuous Tracheal Gas Insufflation (CTGI) reduce the age at the weaning of any ventilatory support and/or oxygen supplementation.

Researchers will compare the clinical outcome of patients mechanically ventilated with the CTGI-device to the outcome of patients ventilated without the CTGI device, to see if the CTGI ventilation works to reduce ventilation dependence.

Participants will:

• Be mechanically ventilated using CTGI (if randomly assigned in the CTGI-group), for the entire endotracheal ventilation period during their stay in the neonatal intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Age at birth between 23 weeks gestation + 0 days and 26 weeks gestation + 6days
* Age between 0 and 7 days of life
* Need for intubation and mechanical ventilation before day 8 of life
* Availability of the Research-associated medical devices
* Beneficiary of a social security system (in France: CMU or securité sociale)
* Parental consent for their infant to participate in this trial

Exclusion Criteria:

* Known Severe Congenital Malformation (potential life-threatening malformation)
* Known Preexisting Severe Intraventricular Haemorrhage (grade 3 or 4) and/or other brain abnormality that can alter life prognosis
* Known Genetic Disorder (potential life-threatening malformation)
* Preexistent mechanical ventilation for a duration of more than 12 hours
* Participation in another interventional research trial before inclusion

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2025-02-13 (Estimated); Primary Completion 2027-04-02 (Estimated); Study Completion 2029-04-03 (Estimated)

PRIMARY OUTCOMES:
Cumulative duration of all periods of non-invasive ventilation | From birth to the end of hospital stay, up to maximum 45 weeks of corrected gestational age.
  The cumulative duration of all periods of non-invasive ventilation, in days, starting from birth, and up to maximum 45 weeks corrected gestational age. Non-invasive ventilation includes all types of positive pressure support non-invasive ventilation and high flow nasal cannula ventilation (HFNC).

SECONDARY OUTCOMES:
Number of participants deceased | From enrollment to the date of the end of the hospital stay, up to maximum 5 months of life
  For each arm: mortality rate during initial hospitalization.
Measure of the Driving Pressure during mechanical ventilation | From enrollment to the date of the end of the hospital stay, up to maximum 5 months of life
  Mean Driving pressure (∆P: Ppeak-PEEP) collected each 12 hours for all patients on invasive mechanical ventilation.
Measure of expiratory tidal volume during mechanical ventilation. | From enrollment to the date of the end of the hospital stay, up to maximum 5 months of life
  Mean expiratory tidal volume (VT) collected each 12 hours for all patients on invasive mechanical ventilation.
Measure of carbon dioxide partial pressure (PCO2) on blood gas | From enrollment up to maximum 15 days of life
  Carbon dioxide partial pressure (PCO2) on patient's blood gas during mechanical ventilation
Measure of Transcutaneous Carbon dioxide partial pressure (TcPCO2) | From enrollment to the date of the end of the hospital stay, up to maximum 5 months of life
  Transcutaneous measure of Carbon dioxide partial pressure (TcPCO2) collected each 12 hours during mechanical ventilation.
Number of participants who received a second dose of surfactant | From birth up to maximum 7 days of life.
  Rates of patients with more than one dose of surfactant replacement therapy.
Number of participants treated with high-frequency ventilation (HFV) or high-frequency oscillatory ventilation (HFOV). | From enrollment to the date of the end of the hospital stay, up to maximum 5 months of life
  Rates of patients treated with High Frequency ventilation (HFV) or High frequency oscillatory ventilation (HFOV) during invasive mechanical ventilation.
Use of Inhaled Nitric Oxide (iNO therapy) | From enrollment to the date of the end of the hospital stay, up to maximum 5 months of life
  Rates of patients treated with nitric oxyde (iNO) during invasive mechanical ventilation.
Number of participant with Severe hypoxemia | From enrollment to the date of the end of the hospital stay, up to maximum 5 months of life
  Rates of patients with Oxygenation Index ≥ 10
Number of participants treated for Pneumothorax | From enrollment to the date of the end of the hospital stay, up to maximum 5 months of life
  Rates of patients with treated Pneumothorax (Needle Thoracentesis or Chest Drainage)
Number of participants treated with Systemic Corticosteroids for Prevention or Management of Bronchopulmonary Dysplasia (BPD) | From enrollment to the date of the end of the hospital stay, up to maximum 5 months of life
  Rates of patients treated with systemic corticosteroids for the prevention or management of BPD and number of days of treatment, excluding prophylactic hydrocortisone treatment in the first 10 days of life.
Number of participants diagnosed as Bronchopulmonary Dysplasia (BPD) | From two days before 36 weeks of corrected gestational age until two days after 36 weeks of corrected gestational age..
  Rates of patients with Bronchopulmonary Dysplasia (BPD) diagnosed at 36 weeks of corrected gestational age.
Number of participants with unplanned extubation | From birth to the date of the end of the hospital stay, up to maximum 5 months of life
  Rates of unplanned extubations per 100 ventilator days, and context.
Calculation of days with invasive mechanical ventilation for each participant. | From birth to the date of the end of the hospital stay, up to maximum 5 months of life
  Number of days spent on invasive mechanical ventilation
Calculation of the mean age at definitive weaning from invasive ventilation for the participants in each arm. | From birth to the date of the end of the hospital stay, up to maximum 5 months of life
  Age at total weaning from invasive mechanical ventilation
Age of participants at definitive weaning from all positive pressure ventilatory support | From birth to the date of the end of the hospital stay, up to maximum 5 months of life
  The age in days when the infant is definitively weaned from invasive and non-invasive positive pressure ventilation, excluding High Flow Nasal Canula (HFNC) and Low Flow Nasal Canula ventilation (LFNC).
Age of the participants at the definitive withdrawal of any Ventilatory Support | From birth to the date of the end of the hospital stay, up to maximum 5 months of life
  The age in days when the infant is definitively weaned from invasive and non-invasive ventilation, including High-Flow Nasal Cannula (HFNC). This excludes Low-Flow Nasal Cannula (LFNC), with or without supplemental oxygen delivery.
Age of the participants at definitive O2 weaning. | From birth to the date of the end of the hospital stay, up to maximum 5 months of life
  The age in days when the patient is definitively weaned from oxygen supplementation. This includes being weaned from any respiratory support system, as well as from Low-Flow Nasal Cannula, with or without supplemental oxygen delivery.
Number of participants with Late-onset primary bloodstream infections | From birth to the date of the end of the hospital stay, up to maximum 5 months of life
  Rates of Late-onset primary bloodstream infections using CDC surveillance definitions, calculated for 1000 central-line days.
Number of participants with Neuroimaging complications | From birth to the date of the end of the hospital stay, up to maximum 5 months of life
  Rates of acquired neuroimaging complications: Periventicular Leucomalacia, Cerebellar haemorrhage, Intra-Ventricular Haemorrhage Grade 3 and 4.
Number of participants Treated for Retinopathy (ROP) | From birth to the date of the end of the hospital stay, up to maximum 5 months of life
  Rates of Retinopathy (ROP) receiving either retinal laser or intravitreal anti-VEGF therapy.
Number of days for each participant of Exposure to systemic analgesic or sedatives treatments | From birth to the date of the end of the hospital stay, up to maximum 5 months of life
  Number of days with systemic analgesic or sedative treatments.
First cytokine dosage in tracheal aspirates. | Between 24 hours to 48 hours of life.
  Mean Cytokines dosage from tracheal aspirates in intubated patients (one unique aspiration). This outcome will be assessed only for patients enrolled in the study and on mechanical ventilation between 24 and 48 hours of life.
Second cytokine dosage in tracheal aspirates. | Between day 4 to day 5 of life.
  Mean Cytokines dosage from tracheal aspirates in intubated patients (one unique aspiration). This outcomes will be assessed only for patients enrolled in the study and on mechanical ventilation between day 4 and 5 of life.
Third cytokine dosage in tracheal aspirates. | Between day 10 to day 12 of life.
  Mean Cytokines dosage from tracheal aspirates in intubated patients. This outcomes will be assessed only for patients enrolled in the study and on mechanical ventilation between day 10 and day 12 of life.
Number of participants requiring hemodynamic support. | From enrollment in the study to the date of the end of the hospital stay, up to maximum 5 months of life
  Rates of patients receiving hemodynamic support during their hospital stay (systemic catecholamines, volume expansion).
Measurement of average weight gain for all study participants in each arm. | From birth to the date of 36 weeks of corrected gestational age.
  Weight gain in grams between birth weight and weight at 36 weeks of corrected gestational age.
Number of days for each participant in the study with central venous line | From birth to the date of the end of the hospital stay, up to maximum 5 months of life
  Addition of all the periods the patients has a central line, in days.
Resuts of Neurodevelopmental Follow-up for surviving participants. | At 2 years of corrected age (± 2 months)
  Results of the validated French version of the "Ages & stages questionnaires" (ASQ3), a developmental screening tool based on parental reporting for their child. This tool will be sent to the parents, and collected.
Number of participants with Cerebral Palsy | At 2 years of corrected age (± 2 months)
  Rates of patients with cerebral palsy.
Number of participants with visual disorders at 2 years of age | At 2 years of corrected age (± 2 months)
  Rates of patients with severe visual disorders defined as a need for glasses at 2 years of corrected age (± 2 months)
Number of participants necessitating respiratory drugs during the two first years of life. | From the date of discharge from the hospital to 2 years of age
  Rates of patients with respiratory symptoms in the first two years, defined as the need for respiratory medications (inhaled or systemic) at any time in this period.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana PATKAI, MD, Principal Investigator — CHU Cochin-Port Royal; Valérie BIRAN, MD, PhD, Principal Investigator — CHU Robert Debré; Cyril FLAMANT, MD, PhD, Principal Investigator — Nantes University Hospital; Fabrice DECOBERT, MD, Principal Investigator — CHI de Créteil
Locations (4):
- France (4):
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Hopistalier Universitaire Cochin Port Royal aphp, Paris
  - Centre hospitalier Robert Debré aphp, Paris

IPD SHARING:
Plan to Share IPD: No